CLINICAL TRIAL: NCT01139736
Title: Manipulation of Visceral Hypersensitivity With Probiotic Bacteria in Irritable Bowel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Dr Siew C Ng, The Chinese Unviersity of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBS Probiotics
Record Dates: First submitted 2010-06-03; First posted 2010-06-09 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2011-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; IBS; probiotics; rectal sensitivity; gut flora; gut bacteria
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Probiotics (Experimental): IBS Patients will receive VSL#3 (450 billion lyophilized bacteria/sachet) twice daily for 4 weeks. VSL#3 was selected for use in this study because (a) it contains three different Bifidobacteria strains (in addition to lactobacilli and streptococci) and the limited evidence available Bifidobacteria as the most effective probiotics in IBS .
  Interventions: Dietary Supplement: VSL#3

INTERVENTIONS:
Dietary Supplement: VSL#3 — IBS Patients will receive VSL#3 (450 billion lyophilized bacteria/sachet) twice daily for 4 weeks

SUMMARY:
Irritable bowel syndrome is a common digestive disorder worldwide. However, there is no effective treatment of irritable bowel syndrome. Visceral pain thresholds in response to stress are lower in patients with IBS compared to healthy volunteers, but the triggers to visceral hypersensitivity remain largely unknown. Animal models suggest roles for both host immune response and intestinal bacteria in the induction of visceral hypersensitivity. For instance colorectal distension increased in association with an alteration in bacterial flora induced by antibiotic therapy, which suggest a relationship between bacterial gut content and visceral afferent processing. Intestinal bacteria play a significant role in inducing IBS. Clinical studies have shown that manipulation of the commensal microbiota with probiotic bacteria, in particularly preparations that contain bifidobacteria, can alleviate IBS symptoms. Serotonin (5-HT) plays a crucial role in the regulation of gastrointestinal physiology and alterations in mucosal serotonin signaling is a possible mechanism of altered function and sensation in patients with IBS. Impairment of serotonin reuptake transporter (SERT) expression and function may also play a role in IBS. The investigators hypothesise that bacteria modulate sensory afferent and serotonin signaling necessary for visceral sensation and that these pathways can be targeted for therapy of IBS using probiotic bacteria. The first part of this study will be a cross-sectional study comparing the colonic microbiota and SERT polymorphisms in IBS patients and healthy controls. The second part will be an open-label pilot study to assess the effects of oral probiotic bacteria in visceral hypersensitivity and mucosal microbiota in patients with IBS. Clinical response will be assessed based on IBS symptom score and rectal sensitivity, and changes in mucosa microbiota will be measured using 454 pyrosequencing. This proposal will provide novel data on gut microbiota in Asian IBS patients, and explore the mechanisms underlying visceral hypersensitivity to direct future targeting of therapy in IBS.

DETAILED DESCRIPTION:
Background

An incomplete understanding of the mechanisms underlying irritable bowel syndrome (IBS) has hampered the development of an effective therapy for this condition. This is long overdue for a condition that affects at least 20 percent of the population (1), and has a major impact on patient's quality of life (QOL) (2).Current understanding of the underlying aetiology and pathogenesis of IBS is centered on two levels: the brain-gut axis which provides concept of how stress, emotion and psychological conditions all alter the perception of IBS symptoms. Within the intestinal wall, the patho-physiological mechanisms that are implicated in IBS include infection, immune activation, dysmotility, abnormal fermentation and visceral hypersensitivity. Studies have shown that visceral pain thresholds in response to stress are lower in patients with IBS compared to healthy volunteers (3). This hypersensitivity is apparent in response to both a physical and chemical stimulus but the triggers to visceral hypersensitivity remain largely unknown. intestinal bacteria play a significant role in inducing IBS. For instance post-infectious IBS developed in a subgroup of patients following a bout of gastroenteritis (4). Manipulation of the commensal microbiota can alleviate IBS symptoms and there is some evidence that probiotic preparations containing certain Bifidobacteria may be particularly effective (5). This proposal will focus on further exploration of the mechanisms underlying visceral hypersensitivity to direct future targeting of therapy with probiotic preparation.

Aims The aims of this study are (i) to identify IBS-associated changes in intestinal microbiota; (ii) to study SERT expression and genotyping, and their relationship with the gut microbiota, and (iii) to determine whether probiotic therapy alters visceral sensitivity in IBS patients and whether probiotic-induced changes in visceral hypersensitivity are associated with changes in the intestinal microbiota.

Hypothesis The investigators postulate that bacteria modulate sensory afferent signalling and serotonin signalling, necessary for visceral sensation and that these pathways can be targeted for therapy of IBS using probiotic bacteria.

RESEARCH PLAN This study consists of two parts. The first part will be a cross-sectional study comparing the colonic microbiota and SERT expression in IBS patients and healthy controls. The second part will involve a pilot open-label study to assess the effects of oral probiotic bacteria in visceral hypersensitivity, SERT expression and mucosal microbiota in patients with IBS.

Baseline visit Ten subjects with IBS will be recruited from outpatient clinics. Disease severity will be determined at enrolment with a validated IBS symptom questionnaire. Routine blood tests including full blood count, biochemistry profile and C-reactive protein will be obtained. Rectal sensitivity to pressure and pain will be assessed with Barostat device. Barostat device has been used in many other studies as a measure of visceral hypersensitivity. Equipment for both tests is currently in use at our laboratory. A baseline colonoscopy will be performed and rectal biopsies will be taken. Ten controls undergoing screening colonoscopy for polyps or colorectal cancer and subsequently found to have a normal colonoscopy will be included to participate in the FGI-Bx study, in which their tissue samples would be used in this study.

Baseline samples from IBS:

1 rectal tissue (formalin fixed for histology) 2 rectal tissues (SERT polymorphism) 3 rectal tissues (mucosal microbiota) 5ml blood in EDTA tube (SERT polymorphism)

Samples from controls:

1 rectal tissue (formalin fixed for histology) 2 rectal tissues (SERT polymorphism) 3 rectal tissues (mucosal microbiota) 5ml blood in EDTA tube (SERT polymorphism)

Intervention IBS Patients will receive VSL#3 (450 billion lyophilized bacteria/sachet) twice daily for 4 weeks. VSL#3 was selected for use in this study because (a) it contains three different Bifidobacteria strains (in addition to lactobacilli and streptococci) and the limited evidence available Bifidobacteria as the most effective probiotics in IBS (13) . A flow chart of the study is in appendix 1.

Week 4 Assessment

Clinical response to probiotic therapy Assessments will be made at baseline and at day 28 of therapy. The three symptoms of IBS will be assessed to determine response to therapy: abdominal pain/ discomfort, bloating/ distension and bowel movements, each scored on an ordinal scale (Likert scale; maximum score 7) and on a 100mm visual analogue scale (VAS; maximum score 100). A composite score with the sums of the 3 cardinal symptoms will also be calculated for each patient (Likert scale maximum score 21) (VAS; maximum score 300). Repeat rectal sensitivity testing will be performed.

Changes in mucosa microbiota in response to probiotic therapy Assessments will be made at baseline and at day 28. Because of the somewhat invasive nature of a repeat colonoscopy, the investigators will only perform a flexible sigmoidoscopy to obtain rectal biopsies after probiotic treatment.

Week 4 samples from IBS:

1. rectal tissue (formalin fixed for histology)
2. rectal tissues (SERT polymorphism)
3. rectal tissues (mucosal microbiota)

5ml blood in EDTA (SERT polymorphism)

Six months follow-up Patients will be contacted at 6 months to reassess symptom scores to determine longer-term impact of therapy.

COLONOSCOPY Colonoscopy will be performed as an outpatient procedure under conscious sedation with intravenous diazepam and pethidine. Subjects will receive bowel preparation with PEG. For flexible sigmoidoscopy, an unprepared examination with be performed and four biopsies will be obtained at 15cm from the anal verge.

RECTAL BAROSTAT The barostat device contains a built-in computer system that can be programmed to automatically perform distensions of balloon with fixed time lags and bag pressure increments. Variation in balloon volume in a constant pressure reflects the change in tone and compliance of the visceral wall. Furthermore, through a programmed variation in intraballoon pressure, the sensory threshold of subject can be evaluated.

The patient is instructed to administer 4.5 fl oz of sodium phosphates rectally 4 hours before study at home for rectal cleansing. After a 3-hour fast, the participant will be positioned in left lateral position. A barostat bag is inserted into the rectum. The barostat device is connected to the barostat catheter using a low compliance PVC tubing.

After 10 minutes of resting, phasic isobaric rectal distensions are performed automatically using ascending method of limits (AML) protocol with successive increments of 4 mm Hg (40-second duration) alternating with intermittent periods of bag deflation (40 seconds). During each distension phase, the participant is requested to report the perception ratings by pressing on the perception panel of barostat device with the following scale: (1) No sensation of balloon distension, (2) the first sensation of balloon distension, (3) desire for defecation, (4) maximum tolerable sensation. The procedure will be stopped when pain or maximum tolerable sensation is reported. The sensory threshold is defined as lower limit of the bag pressure that evokes the first sensation of balloon distension. The pain threshold is defined as pressure that elicits a "pain" response or maximum tolerable sensation.

MUCOSAL MICROBIOTA Colonic samples will be taken to represent adherent bacterial flora. All samples will be stored at -80 degree Celsius until use. Each sample will be added to tubes containing 500µl of phenol: Chloroform: isoamyl alcohol (24:24:1), and 500µl of 0.1mm diameter zirconia/silica beads (Biospec Products, Barthesville, OK). Microbial cells will be disrupted mechanically at 23 degree Celsius with a bead beater (Biospec Products, instrument set on high for 2 minutes). Isolated DNA will be fractionated by electrophoresis through 1% agarose gels, and the dominant band will be purified by MiniElute Gel Extraction kit (Qiagen).

Amplification of the bacterial 16S ribosomal RNA sequences for pyrosequencing will be performed by PCR. For each sample, 100-200mg of purified genomic DNA will be amplified by using primers BSR357-A and BSF8-B, which anneal to conserved regions of bacterial 16s rRNA gene. The PCR products will be sequenced using the 454 Life Sciences Technology Genome Sequencer FLX system (provided by Faculty of Science, CUHK). Quality control will be achieved by the following criteria: the sequence should (i) show a perfect match to the bar code and 16S ribosomal RNA gene primer, (ii) be at least 50 nucleotide in length, (iii) have no more than two undetermined bases in the sequence read, and (iv) have at least a 75% match to a previously determined 16S ribosomal RNA gene sequence. Operational taxonomic unit (OTU) clustering and analysis will be carried out using OTUPicker. Clustering and principal coordinate analysis will be conducted using UniFrac. Since errors in pyrosequencing occur at a rate of only 0.25%, most of the 400-nucleotide sequences that remain after filtering will contain either 0 or 1 error. This level of sequencing error will not affect the taxonomic analysis.

The final data set for colonic microbial taxonomic analysis will be compared with the 1,358,426-sequence Ribosomal Database Project Release 10.

SEROTONIN TRANSPORTER POLYMORPHISM For genotyping, DNA will be isolated from blood platelet (from venous blood) and colon biopsies by standard phenol/chloroform extraction.

The 44-bp insertion/deletion polymorphism in the promoter region (SERT-P) will be analysed by PCR of sample DNA with forward primer 5'-GAG GGA CTG AGC TGG ACA ACC AC-3' and reverse primer 5'-GGC GTT GCC GCT CTG AAT GC-3'. The expected product sizes are 484 bp for deletion (s) and 528 bp for insertion (l) respectively.

The 17-bp VNTR polymorphism of SERT gene intron 2 will be studied by PCR of sample DNA with forward primer 5'-GTC AGT ATC ACA GGC TGC GAG-3' and reverse primer 5'-TGT TCC TAG TCT TAC GCC AGT-3'. The expected product sizes for alleles 9, 10, 11 and 12 are 253bp, 270bp, 287bp and 304bp respectively.

The colonic and platelet SERT protein expressions will also be studied by real time PCR and western blot method.

ELIGIBILITY:
Inclusion Criteria:

Symptoms of abdominal pain or discomfort of at least 3 times a month, in the last 6 months, associated with 2 or more of the following:

* Improvement with defecation
* Onset associated with a change in frequency of stool
* Onset associated with a change in form (appearance) of stool

Exclusion Criteria:

* history of weight loss or rectal bleeding
* history of psychiatric illness (severe depression, mania and schizophrenia)
* history of active infection
* recent antibiotic therapy or anti-inflammatory medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Clinical symptoms | 4 weeks post probiotic

SECONDARY OUTCOMES:
Differences in gut microbiota between IBS patients and controls | 1 year
Difference in gut microbiota post probiotic in IBS patients | 1 year
Differences in blood and mucosal SERT polymorphisms between IBS patients and controls | 1 year
Rectal sensitivity | 4 weeks post probiotics

CONTACTS AND LOCATIONS:
Overall Officials: Siew C Ng, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong